CLINICAL TRIAL: NCT05433532
Title: A Phase Ⅱ, Open Label, Single Arm, Single-Center Study to Evaluate the Efficacy and Safety of Azacitidine，Venetoclax，and Flumatinib in Newly Diagnosed Ph-positive Acute Leukemia and CML-AP/BP Patients
Brief Title: Study of Azacitidine，Venetoclax，and Flumatinib in Newly Diagnosed Ph-positive Acute Leukemia and CML-AP/BP Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AZA+VEN+TKI
Record Dates: First submitted 2022-06-14; First posted 2022-06-27 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Philadelphia Chromosome; Acute Myeloid Leukemia; Acute Lymphoblastic Leukemia; Chronic Myeloid Leukemia; Mixed Phenotype Acute Leukemia
Keywords: Ph-positive AL; CML-AP/BP; Azacitidine+Venetoclax+Flumatinib
MeSH Terms: conditions — Philadelphia Chromosome; Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia, Biphenotypic, Acute | interventions — Azacitidine; venetoclax; flumatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Azacitidine，Venetoclax，and Flumatinib Regimen (Experimental): See Detailed Description.
  Interventions: Drug: Azacitidine; Drug: Venetoclax; Drug: Flumatinib

INTERVENTIONS:
Drug: Azacitidine — Azacitidine: 75mg/m2 qd, d1-d7, subcutaneous injection
Drug: Venetoclax — Venetoclax: 100mg d1, 200mg d2, 300mg d3, 400mg d4-d14 or 21, oral (Adjusted according to the peripheral blood BCR/ABL1 results on day 14)
Drug: Flumatinib — Flumatinib: 600mg qd, d4-d21, oral

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of azacitidine，venetoclax，and flumatinib in newly diagnosed Philadelphia chromosome-positive acute leukemia and accelerated phase or blast phase chronic myeloid leukemia patients.

DETAILED DESCRIPTION:
This is a phase Ⅱ, open-label, single-arm, single-center study in newly diagnosed Ph-positive acute leukemia and CML-AP/BP patients. The patients will receive azacitidine, venetoclax, and flumatinib regimen in the induction treatment. The patients who respond to induction treatment will undergo consolidation treatment, and an optional allogeneic hematopoietic stem cell transplantation and post-transplantation maintenance treatment with induction therapy according to patient's wishes.

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed Ph-positive ALL/AML/MPAL and CML-AP/BP without the history of chemotherapy or target therapy.
2. Age 18-65.
3. Eastern Cooperative Oncology Group (ECOG) score: 0-3.
4. Total serum bilirubin ≤ 2 x upper limit of normal (ULN), alanine aminotransferase (ALT) ≤ 1.5 x ULN, aspartate aminotransferase (AST) ≤ 1.5 x ULN.
5. Creatinine clearance ≥ 30 mL/min.
6. Serum lipase ≤ 1.5 x ULN, amylase =< 1.5 x ULN.
7. No consumption of grapefruit, grapefruit products, Seville oranges, or star fruit within 3 days prior to starting venetoclax.
8. Provide informed consent.

Exclusion Criteria:

1. Patients with another malignant disease.
2. Patients has participated in or participating in other clinical trials.
3. Patients with uncontrolled active infection.
4. Patients with left ventricular ejection fraction < 0.5 by echocardiography or grade III/IV cardiovascular dysfunction according to the New York Heart Association Classification.
5. Patients with HIV infection, active tuberculosis infection, or active hepatitis B or hepatitis C infection.
6. Patients with uncontrolled active bleeding.
7. Patients with history of previous chemotherapy or target therapy (except for oral hydroxyurea and/or leukopheresis for lowering white blood cell counts).
8. Pregnant and lactating women; patients of childbearing potential should be willing to practice methods of contraception throughout the study period.
9. Patients with other commodities that the investigators considered not suitable for the enrollment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2024-04-13 (Actual); Study Completion 2024-04-13 (Actual)

PRIMARY OUTCOMES:
CMR | End of cycle 2 (each cycle is 28 days)
  Complete molecular remission (CMR) was defined as undetectable BCR/ABL transcript.

SECONDARY OUTCOMES:
CR/CRi, MRD-negative CR, CCyR, MMR | End of cycle 1 and 2 (each cycle is 28 days)
  Complete remission (CR) was defined as < 5% bone marrow blasts in an aspirate with spicules and independent of transfusions.
  CR with incomplete hematologic recovery (CRi) was defined as <5% bone marrow blasts, either ANC<1×10^9/L or platelets < 100×10^9/L, transfusion independence but with persistence of cytopenia.
  Minimal residual disease (MRD)-negative CR was defined as a leukemic cell count below the sensitivity threshold of 1×10-4 (0.01%) bone marrow mononuclear cells (MNCs) by multiparameter flow cytometry.
  Complete cytogenetic response (CCyR) was defined as lack of Ph in ≥ 20 bone marrow metaphases.
  Major molecular response (MMR) was defined as a BCR-ABL/ABL transcript ratio of 0.1% (international scale).
Number of adverse events | End of cycle 1 and 2 (each cycle is 28 days)
  Adverse events are evaluated with CTCAE V5.0.
RFS | 2 years
  Relapse-free survival (RFS) was the duration from the day of CR to leukemia relapse, death, or last follow-up.
OS | 2 years
  Overall survival (OS) was the time from enrollment to death for any reason.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaowen Tang, Ph.D, Study Chair — The First Affiliated Hospital of Soochow University
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No